CLINICAL TRIAL: NCT07155174
Title: A Phase 2 Randomized, Open Label, Multicenter Study to Evaluate the Optimal Dose, Safety, and Efficacy of ABBV-706 in Combination With Atezolizumab Versus Standard of Care as First-Line Treatment in Subjects With Previously Untreated Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: A Study to Evaluate the Optimal Dose, Adverse Events and Change in Disease Activity of Intravenous ABBV-706 in Combination With Atezolizumab Versus Standard of Care as First-Line Treatment in Adult Participants With Previously Untreated Extensive Stage Small Cell Lung Cancer
Acronym: SEZanne
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-633; 2024-517490-24 (Other: EU CT)
Record Dates: First submitted 2025-08-28; First posted 2025-09-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; ABBV-706; Etoposide; Carboplatin; Atezolizumab; Lurbinectedin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Etoposide; Carboplatin; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Safety Lead-In: ABBV-706 Dose A (Experimental): Participants will receive ABBV-706 dose A in combination with atezolizumab, as part of the approximately 69.5 month study duration.
  Interventions: Drug: ABBV-706; Drug: Atezolizumab
- Safety Lead-In: ABBV-706 Dose B (Experimental): Participants will receive ABBV-706 dose B in combination with atezolizumab, as part of the approximately 69.5 month study duration.
  Interventions: Drug: ABBV-706; Drug: Atezolizumab
- Safety Lead-In: Stand of Care (SOC) (Experimental): Participants will receive SOC (etoposide, carboplatin, atezolizumab, and optional lurbinectedin), as part of the approximately 69.5 month study duration.
  Interventions: Drug: Atezolizumab; Drug: Etoposide; Drug: Carboplatin; Drug: Lurbinectedin
- Expansion: ABBV-706 Dose A (Experimental): Participants will receive ABBV-706 dose A in combination with atezolizumab, as part of the approximately 69.5 month study duration.
  Interventions: Drug: ABBV-706; Drug: Atezolizumab
- Expansion: ABBV-706 Dose B (Experimental): Participants will receive ABBV-706 dose B in combination with atezolizumab, as part of the approximately 69.5 month study duration.
  Interventions: Drug: ABBV-706; Drug: Atezolizumab
- Expansion: SOC (Experimental): Participants will receive SOC (etoposide, carboplatin, atezolizumab, and optional lurbinectedin), as part of the approximately 69.5 month study duration.
  Interventions: Drug: Atezolizumab; Drug: Etoposide; Drug: Carboplatin; Drug: Lurbinectedin

INTERVENTIONS:
Drug: ABBV-706 — Intravenous (IV) Infusion
  Arms: Expansion: ABBV-706 Dose A; Expansion: ABBV-706 Dose B; Safety Lead-In: ABBV-706 Dose A; Safety Lead-In: ABBV-706 Dose B
Drug: Atezolizumab — IV Infusion
Drug: Etoposide — IV Infusion
  Arms: Expansion: SOC; Safety Lead-In: Stand of Care (SOC)
Drug: Carboplatin — IV Injection
  Arms: Expansion: SOC; Safety Lead-In: Stand of Care (SOC)
Drug: Carboplatin — IV Infusion
  Arms: Expansion: SOC; Safety Lead-In: Stand of Care (SOC)
Drug: Lurbinectedin — IV Infusion
  Arms: Expansion: SOC; Safety Lead-In: Stand of Care (SOC)

SUMMARY:
Small cell lung cancer (SCLC) is characterized by aggressive and rapid growth and a tendency to develop early spread to distant sites including mediastinal lymph nodes, liver, bones, adrenal glands, and brain. The purpose of this study is to assess safety, dose, change in disease activity of ABBV-706 given with atezolizumab, compared to standard of care (SOC) treatment (etoposide, carboplatin, atezolizumab, and optional lurbinectedin).

ABBV-706 is an investigational drug being developed for the treatment of SCLC. There are multiple treatment arms in this study. Participants will either receive ABBV-706 given with atezolizumab, at 1 of 2 doses, or SOC. Approximately 180 adult participants will be enrolled in the study across sites worldwide.

In the safety lead-in, participants with SCLC will receive intravenous (IV) ABBV-706 in 1 of 2 doses with IV atezolizumab, or IV SOC. In the expansion portion of the study, participants with SCLC will receive IV ABBV-706 in 1 of 2 doses with atezolizumab, or IV SOC, until the optimal dose of ABBV-706 is determined. The estimated duration of the study is up to 69.5 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed extensive stage small cell lung cancer (ES-SCLC) requiring treatment with first line therapy.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 during the screening period prior to the first dose of study treatment.
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* Suspected brain metastases at screening should have a computed tomography (CT)/ magnetic resonance imaging (MRI) of the brain prior to study entry.

Exclusion Criteria:

* Have received any kind of treatment for limited stage small cell lung cancer (LS-SCLC).
* Known active/symptomatic central nervous system (CNS) metastases should be excluded.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, or any evidence of active ILD/pneumonitis on screening chest computed tomography (CT) scan should be excluded.
* Have any clinically significant conditions that would adversely affect the participant's participation in the study, and the subject should have a life expectancy of at least 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE)s | Up to 69.5 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Progression-Free Survival (PFS) Based on Investigator Assessment | Up to Approximately 24 Months
  PFS is defined as the time from randomization to the first documentation of radiological progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per investigator or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response (OR) as Measured by Overall Response Rate (ORR) Based on Investigator Assessment | Up to Approximately 24 Months
  OR is defined as participants achieving a best overall response (BOR) of confirmed complete response (CR)/partial response (PR) per RECIST v1.1 as determined by investigator prior to initiation of subsequent anti-cancer therapy. OR will be summarized by ORR, defined as the proportion of subjects achieving OR and will be summarized for each arm with its associated 95% confidence interval (CI).
Duration of Response (DoR) Based on Investigator Assessment | Up to Approximately 24 Months
  DoR is defined as time from the initial response of CR/PR until the first documentation of radiographical PD according to RECIST v1.1 by investigator or death from any cause, whichever occurs first.
Disease Control (DC) Based on Investigator Assessment | Up to Approximately 24 Months
  DC is defined as achieving an OR or stable disease (SD) according to RECIST v1.1 by investigator at any time prior to subsequent anti-cancer therapy.
OS | Up to Approximately 28 Months
  OS, is defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- United States (2):
  - Ocala Oncology Center /ID# 278269, Ocala, Florida
  - Fort Wayne Medical Oncology And Hematology /ID# 277336, Fort Wayne, Indiana
- Israel (5):
  - Meir Medical Center /ID# 277292, Kfar Saba, Central District
  - Assuta Ashdod Medical Center /ID# 276661, Ashdod, Southern District
  - The Chaim Sheba Medical Center /ID# 276660, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 276663, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 276662, Jerusalem
- Japan (4):
  - Shizuoka Cancer Center /ID# 277243, Sunto-gun, Shizuoka
  - Tokyo Metropolitan Komagome Hospital /ID# 277335, Bunkyo Ku, Tokyo
  - National Cancer Center Hospital /ID# 277237, Chuo-Ku, Tokyo
  - Wakayama Medical University Hospital /ID# 277260, Wakayama, Wakayama
- Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 277267, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-633